CLINICAL TRIAL: NCT00291551
Title: Paracor Ventricular Support System: United States Clinical Investigational Plan
Brief Title: Paracor Ventricular Support System (PVSS) for Patients With Heart Failure
Acronym: PEERLESS-HF
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Resources unavailable to continue study follow-up.
Sponsor: Paracor Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102.1
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Placement of the PVSS Implant — Implant is placed on epicardial surface of the heart surrounding both the right and left ventricles, to provide mechanical support to the ventricular walls.
  Other Names: HeartNet; Ventricular support device; Ventricular elastic support therapy

SUMMARY:
This is a limited safety and feasibility study to evaluate the PVSS Introducer and Paracor Ventricular Support System when used to treat patients with heart failure. The implant, which is loaded onto the delivery system, is placed over the epicardial surface of the right and left ventricles.

No formal hypothesis testing will be performed; descriptive statistics will be used to summarize patient outcomes. The results of the study will be used to guide the design and sample size estimation of future studies.

DETAILED DESCRIPTION:
Please refer to brief summary.

ELIGIBILITY:
Inclusion Criteria:

* NYHA functional class II or III
* Best medical therapy
* Ejection fraction <= 35%

Exclusion Criteria:

* Heart measurements too large or small for implant sizes
* Intra-cardiac thrombus
* Restrictive cardiomyopathy
* Not a candidate for sternotomy
* Expected adhesions
* Previous coronary artery bypass graft (CABG)
* Active infection
* Stroke, surgery, or implantable cardioverter defibrillator (ICD) within 3 months
* Myocardial infarction (MI) within 1 month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-01; Primary Completion 2007-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Abraham, MD, Principal Investigator — Ohio State University
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Division of Cardiovascular Disease, Birmingham, Alabama
  - University of Colorado, Health Sciences Center, Denver, Colorado
  - University of Florida, Division of Cardiology, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - BryanLGH Heart Institute, Lincoln, Nebraska
  - The Ohio State University Heart Center, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Methodist Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 investigational sites enrolled 39 subjects between January 2005 and October 2006.
Groups:
- Non-randomized, Single- Arm, Treatment: Paracor Ventricular Support System (PVSS)/HeartNet Ventricular Support System implanted using the Paracor Ventricular Support System (PVSS)/HeartNet Introducer via a left lateral thoracotomy surgical approach.
Period: Overall Study
Arm/Group | Non-randomized, Single- Arm, Treatment
Started | 39
Completed | 26
Not Completed | 13
Not completed — Death | 7
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants] — Measured as Caucasian, Black, of African heritage, and Hispanic
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 35
    More than one race | 0
    Unknown or Not Reported | 1
Etiology [Number; unit: participants]
  Ischemic | 8
  Non-ischemic | 31
Duration of heart failure [Mean (Standard Deviation); unit: years] | 6.9 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Death or Additional Surgical Session at 6 Months
Time Frame: 6 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Non-randomized, Single Arm, Treatment
Number analyzed (Participants) | 39
participants | 4

2. Secondary Outcome: Implant Success (Number of Participants Successfully Implanted)
Description: "Implant success" refers to the ability to successfully deliver a device onto the epicardial surface and leave the device in a satisfactory position.
Time Frame: 1 day
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 39
participants | 38

3. Secondary Outcome: Change in NYHA Functional Class
Description: Change in NYHA functional class between baseline and 6 months. "Maintained" means the participant's functional class remains the same as baseline. "Improved" means the participant's functional class has improved (become lower in number) by at least one class. "Worsened" means the participatn's functional class has deteriorated (become higher in number) by at least one class.
Time Frame: Baseline to 6 months
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 36
participants
  Improved | 20
  Maintained | 13
  Worsened | 3

4. Secondary Outcome: Changes in Left Ventricular Diameters
Description: Mean change in left ventricular end-diastolic diameter (LVEDD) and left ventricular end-systolic diameter (LVESD) from baseline to 6 months (echocardiographic measurements)
Time Frame: Baseline to 6 months
Population: per protocol
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 33
centimeters
  LVEDD (cm) | -0.3 (0.7)
  LVESD (cm) | -0.1 (0.6)

5. Secondary Outcome: Changes in Left Ventricular Volumes
Description: Mean change in left ventricular end-diastolic volume (LVEDv) and left ventricular end-systolic volume (LVESV) from baseline to 6 months (echocardiographic measurements)
Time Frame: Baseline to 6 months
Population: per protocol
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Non-randomized, Single Arm, Treatment
Number analyzed (Participants) | 35
milliliters
  LVEDV (ml) | -31.6 (65.2)
  LVESV (ml) | -29.6 (61.6)

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction
Description: Mean change in left ventricular ejection fraction from baseline to 6 months (echocardiographic measurements)
Time Frame: Baseline to 6 months
Population: per protocol
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Non-randomized, Single Arm, Treatment
Number analyzed (Participants) | 35
Percentage | 1.6 (6.0)

7. Secondary Outcome: Change in Left Ventricular Mass
Description: Mean change in left ventricular mass from baseline to 6 months (echocardiogram measurements)
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Non-randomized, Single Arm, Treatment
Number analyzed (Participants) | 30
grams | -17.6 (55.3)

8. Secondary Outcome: Changes in 6 Minute Walk
Description: Mean change in 6 minute walk distance (meters) between baseline and 6 months
Time Frame: Baseline to 6 months
Population: per protocol
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 34
meters | 71.5 (122.9)

9. Secondary Outcome: Changes in Cardiopulmonary Tests
Description: Mean change in Peak VO2 (ml/kg/min) between baseline and 6 months
Time Frame: Baseline to 6 months
Population: per protocol
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 32
ml/kg/min | 0 (2.8)

10. Secondary Outcome: Mean Changes in Overall Minnesota Living With Heart Failure (MLHF) Quality of Life Questionnaire Score
Description: The MLHF Quality of Life (QOL) Questionnaire evaluates the effects of heart failure on a subject's physical, emotional, social and mental dimensions of quality of life. Each of 21 questions is scored as to how much heart failure has impacted the subject, from 0-no impact to 5-very much (overall score can range from 0 to 105). Prior studies have shown a 10-point improvement (10-point decrease in overall score) correlated with a 1 NYHA class improvement, and 10-point worsening (10-point increase in score) was associated with a higher risk of hospitalization or death.
Time Frame: Baseline to 6 months
Population: per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 34
score on a scale | -15.8 (22.2)

11. Secondary Outcome: Number of Adverse Events
Description: Total adverse events reported prior to study closure
Time Frame: Study duration
Population: per protocol
Measure: Number; unit: events
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 39
events
  Adverse Events | 276
  Serious Adverse Events | 158

12. Secondary Outcome: Number of Participants Who Died
Description: Total number of patient deaths reported prior to study closure
Time Frame: Study duration
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Non-randomized, Single- Arm, Treatment
Number analyzed (Participants) | 39
participants | 7

ADVERSE EVENTS:
Time Frame: 6 years, 3 months (maximum)
Description: Patients followed from enrollment until study termination, death, or withdrawal
Arm/Group | Non-randomized, Single- Arm, Treatment
Serious Adverse Events (participants affected / at risk) | 30/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-randomized, Single- Arm, Treatment (N=39)
General (General disorders) | 19 (28)
Cardiovascular (Cardiac disorders) | 25 (84)
Gastrointestinal (Gastrointestinal disorders) | 2 (2)
Genital-urinary (Renal and urinary disorders) | 1 (2)
Hematology (Blood and lymphatic system disorders) | 4 (5)
Neurology (Nervous system disorders) | 4 (7)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 10 (18)
Renal (Renal and urinary disorders) | 8 (12)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-randomized, Single- Arm, Treatment (N=39)
General (General disorders) | 32 (118)
Cardiovascular (Cardiac disorders) | 29 (66)
Gastrointestinal (Gastrointestinal disorders) | 9 (9)
Genital-urinary (Renal and urinary disorders) | 12 (14)
Hematology (Blood and lymphatic system disorders) | 4 (6)
Neurology (Nervous system disorders) | 7 (8)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 20 (37)
Renal (Renal and urinary disorders) | 15 (18)

LIMITATIONS AND CAVEATS:
Insufficient resources to continue study follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No